CLINICAL TRIAL: NCT04345848
Title: Preventing COVID-19-associated Thrombosis, Coagulopathy and Mortality With Low- and High-dose Anticoagulation: a Multicentric Randomized, Open-label Clinical Trial
Brief Title: Preventing COVID-19 Complications With Low- and High-dose Anticoagulation
Acronym: COVID-HEP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low recruitement
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Marc Blondon, Attending Physician, Angiology, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-00794
Record Dates: First submitted 2020-04-07; First posted 2020-04-15 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: COVID; Sars-CoV2
Keywords: anticoagulation; heparin; thrombosis
MeSH Terms: conditions — Thrombosis | interventions — Enoxaparin; Heparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapeutic anticoagulation (Experimental): Participants will be treated with therapeutic doses of subcutaneous low-molecular-weight heparin (enoxaparin) or intravenous unfractionated heparin, from admission until the end of hospital stay or clinical recovery.
  Interventions: Drug: Enoxaparin
- Prophylactic anticoagulation (Active Comparator): Participants will be treated with prophylactic doses of subcutaneous low-molecular-weight heparin (enoxaparin) or unfractionated heparin, from admission until the end of hospital stay or clinical recovery. If hospitalized in the intensive care unit, they will receive an augmented thromboprophylaxis regimen as standard of care.
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — Two different doses of anticoagulation
  Other Names: Unfractionated heparin

SUMMARY:
The ongoing COVID-19 pandemic affects millions of humans worldwide and has led to thousands of acute medical hospitalizations. There is evidence that hospitalized cases often suffer from an important infection-related coagulopathy and from elevated risks of thrombosis. Anticoagulants may have positive effects here, to reduce the burden of thrombotic disease and the hyperactivity of coagulation, and may also hold beneficial anti-inflammatory effects against sepsis and the development of ARDS.

The investigators hypothesize that high-dose anticoagulants, compared with low-dose anticoagulants, lower the risk of venous and arterial thrombosis, disseminated intravascular coagulation (DIC) and mortality. This open-label controlled trial will randomize hospitalized adults with severe COVID-19 infection to therapeutic anticoagulation vs. thromboprophylaxis during the hospital stay.

ELIGIBILITY:
Inclusion Criteria: adult patient with COVID-19 infections, admitted to:

* an acute non-critical medical ward with admission D-dimer levels >1,000ng/mL, or
* an acute critical ward (ICU, intermediate care unit)

Exclusion Criteria:

* ongoing or planned therapeutic anticoagulation for any other indication
* contra-indication to therapeutic anticoagulation
* hypersensitivity to heparin
* personal history of heparin-induced thrombocytopenia
* suspected or confirmed bacterial endocarditis
* bleeding events or tendency due to a suspected or confirmed hemostatic bleeding disorder
* organic lesion prone to bleeding
* platelet count <50G/L, Hb level <80g/L
* ongoing or recent (<30 days) major bleeding, ischemic stroke, trauma, surgery
* use of dual antiplatelet therapy
* pregnancy
* bodyweight <40kg or >150kg.
* end of life care setting
* unwillingness to consent
* ongoing participation in a COVID-19 randomized clinical trial testing another therapeutic intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
Composite outcome of arterial or venous thrombosis, disseminated intravascular coagulation and all-cause mortality | 30 days
  Risk of arterial or venous thrombosis, disseminated intravascular coagulation and all-cause mortality

SECONDARY OUTCOMES:
Arterial thrombosis | 30 days
  Risk of ischemic stroke, myocardial infarction and/or limb ischemia
Venous thromboembolism | 30 days
  Risk of symptomatic venous thromboembolism or asymptomatic proximal leg deep vein thrombosis
Disseminated intravascular coagulation | 30 days
  Risk of DIC
All-cause mortality | 30 days
  Risk of all-cause mortality
Sepsis-induced coagulopathy | 30 days
  Risk of SIC
Acute respiratory distress syndrome | 30 days
  Risk of ARDS
Durations of hospital stay, ICU stay, ventilation | 30 days
  Number of days with these care processes
Sequential organ failure assessment score | 30 days
  Highest score per participant
Clinical deterioration | 30 days
  Risk of clinical deterioration

OTHER OUTCOMES:
Major bleeding | 30 days
  Risk of ISTH-defined major bleeding
Clinically relevant non-major bleeding | 30 days
  Risk of ISTH-defined CRNMB
Heparin-induced thrombocytopenia | 30 days
  Risk of documented HIT
PaO2/FiO2 index | 30 days
  Measures of PaO2/FiO2 among participants with mechanical ventilation

CONTACTS AND LOCATIONS:
Locations (4):
- Switzerland (4):
  - Geneva University Hospitals, Geneva
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
  - Ospedale Regionale di Locarno, Locarno
  - Hôpital du Valais, Sion

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208
- [Derived] Flumignan RL, Tinoco JDS, Pascoal PI, Areias LL, Cossi MS, Fernandes MI, Costa IK, Souza L, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Prophylactic anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD013739. doi: 10.1002/14651858.CD013739. PMID 33502773
- [Derived] Levi M, Thachil J, Iba T, Levy JH. Coagulation abnormalities and thrombosis in patients with COVID-19. Lancet Haematol. 2020 Jun;7(6):e438-e440. doi: 10.1016/S2352-3026(20)30145-9. Epub 2020 May 11. No abstract available. PMID 32407672